CLINICAL TRIAL: NCT03006198
Title: Tracking Biologics Along the Silk Road
Acronym: HARIR
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Other Study IDs: CR106936; C0168ARA4017 (Other: Janssen Pharmaceutica N.V., Belgium)
Record Dates: First submitted 2016-12-28; First posted 2016-12-30 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Colitis, Ulcerative
MeSH Terms: conditions — Arthritis; Spondylitis; Colitis; Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (5):
- Cohort 1: Rheumatoid Arthritis: Participants with Rheumatoid arthritis as the major disease treated with REMICADE, SIMPONI or STELARA in clinical practice in the emerging regions of North Africa, the Middle East, and Western Asia will be observed for disease characteristics, treatment and outcomes.
- Cohort 2: Ankylosing Spondylitis: Participants with Ankylosing spondylitis as the major disease treated with REMICADE, SIMPONI or STELARA in clinical practice in the emerging regions of North Africa, the Middle East, and Western Asia will be observed for disease characteristics, treatment and outcomes.
- Cohort 3: Psoriatic Arthritis: Participants with Psoriatic arthritis as the major disease treated with REMICADE, SIMPONI or STELARA in clinical practice in the emerging regions of North Africa, the Middle East, and Western Asia will be observed for disease characteristics, treatment and outcomes.
- Cohort 4: Crohn's Disease: Participants with Crohn's disease as the major disease treated with REMICADE, SIMPONI or STELARA in clinical practice in the emerging regions of North Africa, the Middle East, and Western Asia will be observed for disease characteristics, treatment and outcomes.
- Cohort 5: Ulcerative Colitis: Participants with Ulcerative colitis as the major disease treated with REMICADE, SIMPONI or STELARA in clinical practice in the emerging regions of North Africa, the Middle East, and Western Asia will be observed for disease characteristics, treatment and outcomes.

SUMMARY:
The objective of this study is to explore and describe the disease characteristics, treatment and outcomes of participants with rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, Crohn's Disease or ulcerative colitis as the major disease treated with REMICADE, SIMPONI or STELARA in clinical practice in the emerging regions of North Africa, the Middle East, and Western Asia.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a confirmed diagnosis of rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, Crohn's Disease, or ulcerative colitis. A participant can be included for one disease only; participants with multiple diagnoses should be included for their major disease only
* Initiation of treatment with REMICADE, SIMPONI, or STELARA should be planned at the time of enrollment into this observational study (such treatment should be started within 30 days of enrollment)
* Participant must be either treatment-naïve to biologics or have been treated with no more than 2 different biologic agents before enrollment
* Participant must sign a participation agreement/informed consent form (ICF) allowing data collection and source data verification in accordance with local requirements

Exclusion Criteria:

* Participant who have previously received treatment with REMICADE, SIMPONI, or STELARA must not be enrolled if they start the same therapy a second time
* Participant has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 30 days before baseline data collection
* Participant is currently enrolled in an investigational study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with confirmed diagnosis of rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, Crohn's Disease, or ulcerative colitis as their major disease for which they will be treated with REMICADE, SIMPONI, or STELARA within clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving American College of Rheumatology (ACR) 20 Response | Year 2/early withdrawal
  The ACR 20 Response is defined as greater than or equal to (>=) 20 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=20 percent improvement in 3 of following 5 assessments: patient's assessment of pain using Visual Analog Scale (VAS; 0-10 millimeter [mm], 0 mm=no pain and 10 mm=worst possible pain), patient's global assessment of disease activity by using VAS (the scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas. The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and serum C-Reactive Protein (CRP).
Percentage of Participants Achieving American College of Rheumatology (ACR) 50 Response | Year 2/early withdrawal
  The ACR 50 Response is defined as >=50 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=50 percent improvement in 3 of following 5 assessments: patient's assessment of pain using VAS (0-10 mm, 0 mm=no pain and 10 mm=worst possible pain), patient's global assessment of disease activity by using VAS (the scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by HAQ-DI and serum CRP.
Percentage of Participants Achieving American College of Rheumatology (ACR) 70 Response | Year 2/early withdrawal
  The ACR 70 Response is defined as >=70 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=70 percent improvement in 3 of following 5 assessments: patient's assessment of pain using VAS (0-10 mm, 0 mm=no pain and 10 mm=worst possible pain), patient's global assessment of disease activity by using VAS (the scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by HAQ-DI and CRP.
Percentage of Participants Achieving Assessment of SpondyloArthritis International Society (ASAS) 20 Response | Year 2/early withdrawal
  The ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) participants in 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 20 = 20 percent improvement from baseline and an absolute change >= 10 units on a 0-10 scale (0=no disease activity; 10=high disease activity) for >= 3 domains, and no worsening in remaining domain.
Percentage of Participants Achieving ASAS 40 Response | Year 2/early withdrawal
  The ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) participants in 4 domains: participant global assessment of disease activity, pain, function, inflammation. The ASAS 40 = 40 percent improvement from baseline and an absolute change >= 20 units on a 0-10 scale (0=no disease activity, 10=high disease activity) for >= 3 domains, and no worsening in remaining domain.
Percentage of Participants Achieving ASAS 5/6 Response | Year 2/early withdrawal
  ASAS 5/6 response is a validated composite assessment, reflecting the proportion of treated patients who achieve within a defined timeframe at least 20 percent improvement in score in at least 5 of a conventional set of 6 clinical domains relevant to AS and no worsening in the remaining domain.
Number of Participants With Clinical Response as Assessed by Crohn's Disease Activity Index (CDAI) | Year 2/early withdrawal
  The CDAI will be assessed by collecting information on 8 different Crohn's disease-related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being. The last 4 variables are scored over 7 days by the participant on a diary card. Clinical response defined as reduction of greater than or equal to 70 points and/or 25 percent from baseline in CDAI.
Number of Participants With Clinical Remission as Assessed by CDAI | Year 2/early withdrawal
  The CDAI will be assessed by collecting information on 8 different Crohn's disease-related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being. The last 4 variables are scored over 7 days by the participant on a diary card. Remission will be defined as CDAI less than (<) 150 points.
Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Score for Crohn's Disease | Baseline, Year 2/early withdrawal
  The IBDQ is a 32-item questionnaire used to assess quality of life in participants with inflammatory bowel diseases. Each question has graded responses from 1 (worst situation) to 7 (best situation). Total score ranges from 32 (worst) to 224 (best). Higher scores indicate better quality of life.
Number of Participants With Clinical Response as Assessed by Mayo Score | Year 2/early withdrawal
  Clinical response is defined as a decrease from baseline in the Mayo score by greater than or equal to 30 percent and >= 3 points, and a decrease from baseline in the rectal bleeding sub score to 0 or 1. The Mayo score consists of 4 sub scores (stool frequency, rectal bleeding, endoscopy findings, and physician's global assessment), rated as 0 (normal) to 3 (severe). Total score is calculated as the sum of 4 sub scores and values range from 0 to 12 scores, where 3 to 5 = mild; 6 to 10 = moderate; and 11 to 12 = severe. Higher scores indicate worsening of the disease.
Number of Participants With Clinical Remission as Assessed by Mayo Score | Year 2/early withdrawal
  Clinical remission is defined as a Mayo score less than or equal to 2 points, with no individual sub score greater than 1. The Mayo score consists of 4 sub scores (stool frequency, rectal bleeding, endoscopy findings, and physician's global assessment), rated as 0 (normal) to 3 (severe). Total score is calculated as the sum of 4 sub scores and values range from 0 to 12 scores, where 3 to 5 = mild; 6 to 10 = moderate; and 11 to 12 = severe. Higher scores indicate worsening of the disease.
Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Score for Ulcerative Colitis | Year 2/early withdrawal
  The IBDQ is a 32-item questionnaire used to assess quality of life in participants with inflammatory bowel diseases. Each question has graded responses from 1 (worst situation) to 7 (best situation). Total score ranges from 32 (worst) to 224 (best). Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (8):
- Algiers, Algeria
- Egypt (2):
  - Alexandria
  - Cairo
- Kuwait (2):
  - Hawalli Area
  - Kuwait City
- Doha, Qatar
- Saudi Arabia (2):
  - Mecca
  - Riyadh